CLINICAL TRIAL: NCT00696436
Title: A Double-Blind, Randomized, Placebo-Controlled, 5-Arm Titration Study to Evaluate the Efficacy and Safety of TAK-491 When Compared With Valsartan and Olmesartan in Subjects With Essential Hypertension
Brief Title: An Efficacy and Safety Study of Azilsartan Medoxomil Compared to Valsartan and Olmesartan in Participants With Essential Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-491-019; U1111-1113-9161 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Cardiovascular Disease; High Blood Pressure; Drug Therapy
MeSH Terms: conditions — Hypertension; Essential Hypertension; Cardiovascular Diseases | interventions — azilsartan medoxomil; azilsartan; Valsartan; olmesartan; Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Azilsartan Medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan Medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Valsartan 320 mg QD (Active Comparator)
  Interventions: Drug: Valsartan
- Olmesartan 40 mg QD (Active Comparator)
  Interventions: Drug: Olmesartan
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan medoxomil — Azilsartan medoxomil 20 mg, tablets and matching placebo comparator orally once daily for two weeks.
  Increased to azilsartan medoxomil 40 mg tablets and matching placebo comparator orally, once daily for up to four weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan medoxomil — Azilsartan medoxomil 40 mg, tablets and matching placebo comparator orally, once daily for two weeks.
  Increased to Azilsartan medoxomil 80 mg, tablets and matching placebo comparator orally, once daily for up to four weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD
Drug: Valsartan — Valsartan 160 mg, tablets, and matching placebo comparator orally, once daily for two weeks.
  Increased to Valsartan 320 mg, tablets, and matching placebo comparator, orally, once daily for up to four weeks.
  Other Names: Diovan®
  Arms: Valsartan 320 mg QD
Drug: Olmesartan — Olmesartan 20 mg, tablets and matching placebo comparator, orally, once daily for two weeks.
  Increased to Olmesartan 40 mg, tablets and matching placebo comparator, orally, once daily for up to four weeks.
  Other Names: Benicar®
  Arms: Olmesartan 40 mg QD
Drug: Placebo — Matching placebo, orally, once daily for up to six weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of azilsartan medoxomil, once daily (QD), compared to placebo, valsartan and olmesartan in participants with essential hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled: only about one-third of patients successfully maintain control.

A major component of blood pressure regulation is the renin-angiotensin-aldosterone system. This is a system of hormone-mediated feedback interactions that result in the relaxation or constriction of blood vessels in response to various stimuli. Angiotensin II, a polypeptide hormone, is formed from angiotensin I in a reaction catalyzed by angiotensin-converting enzyme as part of the renin-angiotensin-aldosterone system. Angiotensin II is the principal pressor agent of the renin-angiotensin-aldosterone system and has multiple effects on the cardiovascular system and on electrolyte homeostasis.

TAK-491 (azilsartan medoxomil) is an angiotensin II type 1 receptor antagonist currently being tested as a treatment for essential hypertension.

Study participation is anticipated to be about 10 weeks. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations, electrocardiograms and ambulatory blood pressure monitoring. Outside of the study center, participants will be required wear an ambulatory blood pressure monitoring device at 24 hour intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension (sitting systolic blood pressure between 150 and 180 mm Hg, inclusive, at Day -1 and 24-hour mean systolic blood pressure between 130 and 170 mm Hg, inclusive, at Day 1).
2. Capable of understanding and complying with protocol requirements.
3. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study
4. Clinical laboratory evaluations within the reference range for the testing laboratory or the results are deemed not clinically significant for inclusion into this study by the investigator.
5. Willing to discontinue current antihypertensive medications at Screening Day 21 visit. If the participant is on amlodipine prior to Screening, the participant is willing to discontinue this medication at Screening Day -28.

Exclusion Criteria:

1. Sitting diastolic blood pressure greater than 114 mm Hg at Day -1 (day prior to Randomization).
2. Baseline 24-hour ambulatory blood pressure monitor reading of insufficient quality.
3. Taking or expected to take an excluded medication as described in the Excluded Medications.
4. Hypersensitive to angiotensin II receptor blockers.
5. History of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
6. Clinically significant cardiac conduction defects.
7. Hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
8. Secondary hypertension of any etiology.
9. Noncompliant (less than 70% or greater than 130%) with study medication during run-in period.
10. Moderate to severe renal dysfunction or disease.
11. Known or suspected unilateral or bilateral renal artery stenosis.
12. History of drug or alcohol abuse within the past 2 years.
13. Previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those participants with basal cell or stage I squamous cell carcinoma of the skin).
14. Type 1 or poorly-controlled type 2 diabetes mellitus (glycosylate hemoglobin greater than 8.0%) at Screening.
15. Hyperkalemia as defined by the central laboratory normal reference range at Screening.
16. Alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice at Screening.
17. Upper arm circumference less than 24 cm or greater than 42 cm.
18. Works night (3rd) shift (defined as 11 PM [2300] to 7 AM [0700]).
19. Unwilling or unable to comply with the protocol or scheduled appointments.
20. Currently is participating in another investigational study or has participated in an investigational study within 30 days prior to Randomization.
21. Any other serious disease or condition at Screening or Randomization that would compromise participant's safety, might affect life expectancy, or make it difficult to successfully manage and follow the subject according to the protocol.
22. Has been randomized in a previous azilsartan medoxomil study.
23. Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1291 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (131):
- United States (86):
  - Alabaster, Alabama
  - Ozark, Alabama
  - Green Valley, Arizona
  - Litchfield Park, Arizona
  - Mesa, Arizona
  - Tempe, Arizona
  - Carmichael, California
  - Chula Vista, California
  - Lincoln, California
  - Mission Viejo, California
  - National City, California
  - Pasadena, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - San Dimas, California
  - San Francisco, California
  - San Ramon, California
  - Santa Ana, California
  - Vista, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Littleton, Colorado
  - Longmont, Colorado
  - Cape Coral, Florida
  - Clearwater, Florida
  - Largo, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Palm Harbor, Florida
  - Tallahassee, Florida
  - Dunwoody, Georgia
  - Roswell, Georgia
  - Arlington Heights, Illinois
  - Belleville, Illinois
  - Champaign, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - Vernon Hills, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Terre Haute, Indiana
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Shawnee, Kansas
  - Biddeford, Maine
  - Norwood, Maine
  - Baltimore, Maryland
  - Towson, Maryland
  - Brooklyn Center, Minnesota
  - Chesterfield, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Margate City, New Jersey
  - Glens Falls, New York
  - Great Neck, New York
  - New Hyde Park, New York
  - New Windsor, New York
  - New York, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Columbus, Ohio
  - Norman, Oklahoma
  - Tulsa, Oklahoma
  - Yukon, Oklahoma
  - Ashland, Oregon
  - Eugene, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Tipton, Pennsylvania
  - Charleston, South Carolina
  - Murrells Inlet, South Carolina
  - North Charleston, South Carolina
  - Cleveland, Tennessee
  - Bedford, Texas
  - Dallas, Texas
  - Houston, Texas
  - Missouri City, Texas
  - San Antonio, Texas
  - Sugarland, Texas
  - Tacoma, Washington
- Argentina (14):
  - Carlos Paz, Córdoba Province
  - Córdoba, Córdoba Province
  - Guaymayen, Mendoza Province
  - Bahía Blanca
  - Berazategui
  - Buenos Aires
  - Corrientes
  - Haedo Pcia. de Buenos Aires
  - La Plata
  - Ramos Mejía Pcia. de Buenos Aires
  - Rosario
  - Salta
  - San Miguel de Tucumán
  - San Salvador de Jujuy
- Brazil (9):
  - Belo Horizonte
  - Campinas
  - Fortaleza
  - Goiaenia
  - Joildille
  - Porto Alegre
  - Rio Janeiro
  - São Paulo
  - Sorocava
- Mexico (10):
  - Aguascalientes, Aguascalientes
  - Chihuahua City, Chihuahua
  - Tijuana, Estado de Baja California
  - León, Guanajuato
  - Guadalajara, Jalapa
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosí
  - Xalapa, Veracruz
  - Mexico City
  - Querètaro
- Peru (6):
  - Arequipa
  - Cusco
  - Huaura
  - Ica
  - Lima
  - Trujillo
- Puerto Rico (6):
  - Aguas Buenas
  - Carolina
  - Jardines de Loiza
  - Orocovis
  - Ponce
  - San Juan

REFERENCES:
- [Result] White WB, Weber MA, Sica D, Bakris GL, Perez A, Cao C, Kupfer S. Effects of the angiotensin receptor blocker azilsartan medoxomil versus olmesartan and valsartan on ambulatory and clinic blood pressure in patients with stages 1 and 2 hypertension. Hypertension. 2011 Mar;57(3):413-20. doi: 10.1161/HYPERTENSIONAHA.110.163402. Epub 2011 Jan 31. PMID 21282560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 141 investigative sites in Guatemala, Mexico, Peru, Puerto Rico and the United States from 02 April 2008 to 19 August 2009.
Pre-assignment Details: Participants with essential hypertension were enrolled in one of five, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 20 mg, tablets and matching placebo comparator orally once daily for two weeks.
  Increased to azilsartan medoxomil 40 mg tablets and matching placebo comparator orally, once daily for up to four weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 40 mg, tablets and matching placebo comparator orally, once daily for two weeks.
  Increased to Azilsartan medoxomil 80 mg, tablets and matching placebo comparator orally, once daily for up to four weeks.
- Valsartan 320 mg QD: Valsartan 160 mg, tablets, and matching placebo comparator orally, once daily for two weeks.
  Increased to Valsartan 320 mg, tablets, and matching placebo comparator, orally, once daily for up to four weeks.
- Olmesartan 40 mg QD: Olmesartan 20 mg, tablets and matching placebo comparator, orally, once daily for two weeks.
  Increased to Olmesartan 40 mg, tablets and matching placebo comparator, orally, once daily for up to four weeks.
- Placebo QD: Matching placebo, orally, once daily for up to six weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Started | 280 (Randomized participants only.) | 285 (Randomized participants only. One participant treated but not randomized and is not included.) | 282 (Randomized participants only.) | 290 (Randomized participants only.) | 154 (Randomized participants only.)
Completed | 257 | 255 | 254 | 268 | 141
Not Completed | 23 | 30 | 28 | 22 | 13
Not completed — Adverse Event | 7 | 9 | 8 | 6 | 4
Not completed — Protocol Violation | 3 | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 6 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 4 | 11 | 5 | 7 | 1
Not completed — Lack of Efficacy | 3 | 1 | 5 | 2 | 4
Not completed — Participant Unavailability | 2 | 0 | 2 | 1 | 0
Not completed — Administrative Error | 2 | 0 | 2 | 0 | 0
Not completed — Participant Non-compliance | 0 | 0 | 1 | 2 | 0
Not completed — Administrative Decision | 1 | 0 | 0 | 0 | 0
Not completed — Missing | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD | Total
Number analyzed (Participants) | 280 | 285 | 282 | 290 | 154 | 1291
Age Categorical [Number; unit: participants]
  <45 years | 41 | 38 | 56 | 39 | 20 | 194
  Between 45 and 64 years | 170 | 184 | 178 | 185 | 98 | 815
  ≥65 years | 69 | 63 | 48 | 66 | 36 | 282
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 134 | 130 | 131 | 64 | 592
  Male | 147 | 151 | 152 | 159 | 90 | 699

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -13.42 (0.690) | -14.53 (0.702) | -10.22 (0.696) | -11.99 (0.666) | -0.25 (0.917)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with treatment as a factor and baseline value as a covariate. Unadjusted p-value was presented. Overall 0.05 level of significance for multiple comparisons was controlled using stepwise testing procedure; Mean Difference (Final Values) = -14.27, 95% CI 2-sided [-16.54 to -12.01]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.16, 95% CI 2-sided [-15.41 to -10.91]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.54, 95% CI 2-sided [-4.44 to -0.64]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.31, 95% CI 2-sided [-6.25 to -2.37]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.136, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.43, 95% CI 2-sided [-3.31 to 0.45]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-5.12 to -1.27]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure.
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 6 relative to baseline.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 269 | 270 | 271 | 283 | 148
mmHg | -16.38 (0.959) | -16.74 (0.957) | -11.31 (0.955) | -13.20 (0.935) | -1.83 (1.293)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.92, 95% CI 2-sided [-18.07 to -11.76]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.55, 95% CI 2-sided [-17.71 to -11.40]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.54, 95% CI 2-sided [-6.17 to -0.92]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.43, 95% CI 2-sided [-8.09 to -2.78]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.18, 95% CI 2-sided [-5.81 to -0.55]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.07, 95% CI 2-sided [-7.73 to -2.42]

3. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -8.65 (0.472) | -9.43 (0.480) | -7.09 (0.476) | -7.74 (0.456) | -0.07 (0.627)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with treatment as a factor and baseline value as a covariate. Unadjusted p-value was presented; Mean Difference (Final Values) = -9.36, 95% CI 2-sided [-10.91 to -7.81]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.58, 95% CI 2-sided [-10.12 to -7.04]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.011, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-2.99 to -0.40]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-3.67 to -1.02]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.166, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-2.19 to 0.38]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.020, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-2.88 to -0.24]

4. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 6 relative to baseline.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 269 | 270 | 271 | 283 | 148
mmHg | -6.97 (0.552) | -8.27 (0.551) | -5.11 (0.550) | -6.10 (0.538) | -0.76 (0.744)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.51, 95% CI 2-sided [-9.33 to -5.69]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -6.21, 95% CI 2-sided [-8.03 to -4.39]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.18, 95% CI 2-sided [-3.69 to -0.67]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.17, 95% CI 2-sided [-4.69 to -1.64]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.257, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-2.39 to 0.64]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.86, 95% CI 2-sided [-3.39 to -0.33]

5. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -13.73 (0.724) | -15.02 (0.736) | -10.26 (0.730) | -12.16 (0.699) | -0.11 (0.963)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -14.92, 95% CI 2-sided [-17.30 to -12.54]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -13.63, 95% CI 2-sided [-15.99 to -11.27]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.86, 95% CI 2-sided [-4.85 to -0.87]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.76, 95% CI 2-sided [-6.80 to -2.73]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.119, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-3.55 to 0.40]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.47, 95% CI 2-sided [-5.49 to -1.45]

6. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -8.96 (0.510) | -9.80 (0.518) | -7.23 (0.514) | -7.82 (0.492) | 0.01 (0.677)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.81, 95% CI 2-sided [-11.48 to -8.13]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.96, 95% CI 2-sided [-10.63 to -7.30]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.99, 95% CI 2-sided [-3.39 to -0.58]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.57, 95% CI 2-sided [-4.00 to -1.14]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.107, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.14, 95% CI 2-sided [-2.53 to 0.25]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-3.15 to -0.30]

7. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -12.28 (0.778) | -13.32 (0.792) | -9.66 (0.784) | -11.90 (0.752) | -0.31 (1.035)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -13.00, 95% CI 2-sided [-15.56 to -10.45]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.97, 95% CI 2-sided [-14.51 to -9.43]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.194, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-3.56 to 0.72]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.65, 95% CI 2-sided [-5.84 to -1.46]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.720, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-2.51 to 1.73]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.62, 95% CI 2-sided [-4.79 to -0.45]

8. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -7.65 (0.540) | -8.54 (0.550) | -6.26 (0.544) | -7.82 (0.522) | 0.10 (0.718)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.64, 95% CI 2-sided [-10.42 to -6.87]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.75, 95% CI 2-sided [-9.52 to -5.99]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.341, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-2.21 to 0.77]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.28, 95% CI 2-sided [-3.80 to -0.76]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.821, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-1.30 to 1.64]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.071, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.39, 95% CI 2-sided [-2.89 to 0.12]

9. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -14.03 (0.764) | -15.55 (0.777) | -10.44 (0.770) | -12.23 (0.738) | -0.10 (1.016)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -15.45, 95% CI 2-sided [-17.96 to -12.94]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -13.93, 95% CI 2-sided [-16.42 to -11.43]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-5.42 to -1.22]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.11, 95% CI 2-sided [-7.26 to -2.97]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.091, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-3.88 to 0.29]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.59, 95% CI 2-sided [-5.72 to -1.46]

10. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 237 | 229 | 234 | 254 | 134
mmHg | -9.16 (0.542) | -10.13 (0.551) | -7.42 (0.547) | -7.82 (0.524) | 0.01 (0.721)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -10.14, 95% CI 2-sided [-11.92 to -8.36]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -9.17, 95% CI 2-sided [-10.94 to -7.40]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-3.81 to -0.82]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-4.24 to -1.19]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.076, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.82 to 0.14]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.024, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-3.25 to -0.22]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 236 | 229 | 234 | 254 | 134
mmHg | -12.46 (0.860) | -13.38 (0.873) | -9.14 (0.865) | -11.65 (0.829) | -0.55 (1.142)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -12.84, 95% CI 2-sided [-15.66 to -10.02]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -11.91, 95% CI 2-sided [-14.72 to -9.11]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.149, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.74, 95% CI 2-sided [-4.10 to 0.62]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.24, 95% CI 2-sided [-6.65 to -1.83]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.494, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-3.16 to 1.53]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.007, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-5.72 to -0.93]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 236 | 229 | 234 | 254 | 134
mmHg | -8.69 (0.648) | -8.61 (0.657) | -6.22 (0.651) | -8.25 (0.624) | -0.69 (0.859)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.91, 95% CI 2-sided [-10.03 to -5.79]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.99, 95% CI 2-sided [-10.10 to -5.88]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.691, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-2.14 to 1.42]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.010, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.39, 95% CI 2-sided [-4.20 to -0.57]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.625, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-2.20 to 1.32]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.46, 95% CI 2-sided [-4.27 to -0.66]

13. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as < 140 mm Hg and/or Reduction From Baseline ≥ 20 mm Hg
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 6, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 269 | 270 | 271 | 283 | 148
percentage of participants | 56.5 | 57.8 | 48.7 | 48.8 | 22.3
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for systolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value was presented; Odds Ratio (OR) = 4.98, 95% CI 2-sided [3.15 to 7.88]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.66, 95% CI 2-sided [2.94 to 7.37]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.032, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.03 to 2.03]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.029, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.04 to 2.06]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.080, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.96 to 1.89]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.071, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.97 to 1.92]

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as < 90 mm Hg and/or Reduction From Baseline ≥ 10 mm Hg
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 269 | 270 | 271 | 283 | 148
percentage of participants | 68.8 | 71.1 | 63.8 | 68.2 | 43.9
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for response criteria for diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic diastolic blood pressure as a covariate. The unadjusted p-value was presented; Odds Ratio (OR) = 3.29, 95% CI 2-sided [2.10 to 5.15]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.86 to 4.54]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.306, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.83 to 1.80]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.132, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.92 to 1.97]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.695, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.74 to 1.58]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.381, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.81 to 1.74]

15. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Diastolic and Systolic Blood Pressure Response
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the 3 sitting blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Number analyzed (Participants) | 269 | 270 | 271 | 283 | 148
percentage of participants | 49.1 | 52.6 | 43.9 | 44.5 | 18.2
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-value for joint response criteria for systolic blood pressure and diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value was presented; Odds Ratio (OR) = 5.18, 95% CI 2-sided [3.20 to 8.41]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 4.43, 95% CI 2-sided [2.73 to 7.19]
Statistical Analysis 3: Comparison: Azilsartan Medoxomil 80 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.056, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.99 to 1.94]
Statistical Analysis 4: Comparison: Azilsartan Medoxomil 80 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.036, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.02 to 2.02]
Statistical Analysis 5: Comparison: Azilsartan Medoxomil 40 mg QD vs Olmesartan 40 mg QD; Test type: Superiority or Other; p = 0.317, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.85 to 1.66]
Statistical Analysis 6: Comparison: Azilsartan Medoxomil 40 mg QD vs Valsartan 320 mg QD; Test type: Superiority or Other; p = 0.234, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.87 to 1.73]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Valsartan 320 mg QD | Olmesartan 40 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 2/280 | 3/284 | 3/277 | 4/290 | 2/155
Other Adverse Events (participants affected / at risk) | 18/280 | 12/284 | 21/277 | 23/290 | 14/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=280) | Azilsartan Medoxomil 80 mg QD (N=284) | Valsartan 320 mg QD (N=277) | Olmesartan 40 mg QD (N=290) | Placebo QD (N=155)
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=280) | Azilsartan Medoxomil 80 mg QD (N=284) | Valsartan 320 mg QD (N=277) | Olmesartan 40 mg QD (N=290) | Placebo QD (N=155)
Headache (Nervous system disorders) | 18 | 12 | 21 | 23 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.